CLINICAL TRIAL: NCT05454865
Title: The Effect of Jin Si Herbal Tea on Cancer-related Fatigue of Gynecological Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB110-253-A
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cancer-related Fatigue; Gynecologic Cancer

STUDY DESIGN:
Intervention Model Description: Patients with advanced cancer and moderate to severe cancer-related fatigue were randomized to receive either Jin Si Herbal Tea or a placebo (mimic fluid) for the first treatment cycle (three weeks) in a double-blind manner. On the next cycle (three weeks), all patients received open-label treatment with Jin Si Herbal Tea.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind setting
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jin Si Herbal Tea (Experimental): Jin Si Herbal Tea 1 pack (15 ml) oral use twice daily for two cycles (1 cycle = 3 wks)
  Interventions: Dietary Supplement: Jin Si Herbal Tea
- Placebo group (Placebo Comparator): Mimic Tea 1 pack (15ml) oral use twice daily in the first cycle, using Jin Si Herbal Tea in the 2nd cycle
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Jin Si Herbal Tea — Jin Si Herbal Tea 1 pack PO bid for 2 treatment cycles (1 cycle = 3 weeks)
  Arms: Jin Si Herbal Tea
Dietary Supplement: Placebo — Placebo 1 1pack PO bid for 1 treatment cycle (1 cycle = 3 weeks) and followed by Jin Si Herbal Tea 1 pack PO bid for the 2nd treatment cycle
  Arms: Placebo group

SUMMARY:
Cancer-related fatigue caused by cancer and treatment reduces patients' compliance with treatment. Fatigue caused by chemotherapy usually has multifaceted symptoms, such as being very tired, feeling weak, desperate for rest, or decreased activity. Cancer-related fatigue is often the main reason why patients are reluctant to continue treatment. Even after finished chemotherapy, most patients still feel fatigued.

Therefore, how to solve the patient's fatigue caused by cancer and treatment is a very important issue, and there is no effective treatment at present. This project plans to use the Jin Si herbal tea developed by our hospital to improve cancer-related fatigue.

DETAILED DESCRIPTION:
Cancer-related fatigue caused by cancer and treatment reduces patients' compliance with treatment. Fatigue caused by chemotherapy usually has multifaceted symptoms, such as being very tired, feeling weak, desperate for rest, or decreased activity. Cancer-related fatigue is often the main reason why patients are reluctant to continue treatment. Even after finished chemotherapy, most patients still feel fatigued.

Therefore, how to solve the patient's fatigue caused by cancer and treatment is a very important issue, and there is no effective treatment at present. This project plans to use the Jin Si herbal tea developed by our hospital to improve cancer-related fatigue.

Jin Si Herbal Tea Brief mechanism of action: It contains eight kinds of traditional Chinese medicines, mainly including wormwood, fish needle grass, Ophiopogon japonicas, houttuynia cordata, platycodon, licorice, perilla leaves, and chrysanthemum, which promote lung health including dampness and clean lung heat, diuresis, generate body heat, anti-cold, clean blood, and reduce phlegm.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received chemotherapy
* Patients who understand the experimental process

Exclusion Criteria:

* Unconscious
* Severe disease, not well-controlled patients judged by PI
* Pregnancy, breastfeeding, menstruation during screening phase
* Weakness, allergy to Herbal tea, frequently felt cold

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Brief Fatigue Inventory-Taiwanese (BFI-T) | 2 months
  scores 0-90, higher scores mean the worse outcome
Functional Assessment of Cancer Therapy-General (FACT-G7, Version 4) | 2 months
  scores 0-28, higher scores mean the worse outcome

SECONDARY OUTCOMES:
Laboratory assessment (White Blood Cells count, Differential count) | 2 months
  monitor bone marrow function

CONTACTS AND LOCATIONS:
Overall Officials: DAH-CHING DING, MD, PhD, Principal Investigator — Buddhist Tzu Chi Hospital
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: No